CLINICAL TRIAL: NCT03539380
Title: TRx0237 for the Treatment of Early and Mild-Moderate Alzheimer's Disease: Intermediate-Size Patient Population
Brief Title: TRx0237 for the Treatment of Early and Mild-Moderate Alzheimer's Disease
Status: Available | Type: Expanded Access
Sponsor: TauRx Therapeutics Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: TRx-237-040
Record Dates: First submitted 2018-05-15; First posted 2018-05-29 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — hydromethylthionine

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: TRx0237 — Starting dose of TRx0237 16 mg/day (unless enrolled under earlier version of protocol and are on an established dose), with flexible dosing after 3 months (4-16 mg/day)

SUMMARY:
This is an expanded access program (EAP) for eligible participants. This program is designed to provide continued access to TRx0237 to individual patients with early and mild-moderate Alzheimer's disease who do not qualify for participation in an ongoing clinical trial. Eligible participants must have previously completed participation in a clinical trial of TRx0237 conducted by TauRx or have previously taken TRx0237 in a compassionate use program, among other criteria. Patients will be considered where a physician can demonstrate clinical benefit for a patient not meeting these criteria; in these cases, TauRx will consider participation of the patient on a case-by-case basis.

ELIGIBILITY:
Inclusion Criteria:

* Early (encompassing Mild Cognitive Impairment) or mild to moderate Alzheimer's disease, as confirmed by a cognitive assessment
* Clinical benefit of continued access to TRx0237 is expected to outweigh any perceived risk
* Ability to travel to the named clinic for regularly scheduled visits.
* The patient and/or his/her legal representative have been informed of the potential risks and obligations and have given written informed consent for continued treatment consistent with local requirements.
* Not participating in a clinical trial of another investigational drug.
* Has one (or more) identified adult study partner who either lives with the subject or has sufficient contact to provide assessment of changes in subject behavior and function over time and information on safety and tolerability; is willing to provide written informed consent for his/her own participation; is able to read, understand, and speak the designated language at the study site; agrees to accompany the subject to each study visit
* A female patient of child-bearing potential must use adequate birth control (as defined by the protocol) for at least 90 days before beginning treatment and agree to continue its use whilst on treatment and for 30 days after the last dose of TRx0237.

Exclusion Criteria:

* Swallowing difficulties which prevent taking the medication whole as instructed.
* Unable to comply with this study protocol or has health concerns that may increase risk, in the opinion of the treating physician
* Enrolled in a previous TRx0237 clinical trial and either did not complete the clinical trial, had a significant treatment-related adverse event that could cause an undue risk, or progressed to severe Alzheimer's disease
* Use of drugs for which there is a warning or precaution in the labeling about methemoglobinemia at approved doses (e.g., dapsone, local anesthetics such as benzocaine used chronically, primaquine and related antimalarials)
* Use of clozapine
* Clinically significant cardiovascular disease
* Clinically significant respiratory failure
* History of clinically significant hematological abnormality or hemoglobin value (confirmed upon repeat) below age/sex appropriate laboratory lower limit of normal
* Creatinine clearance <15 mL/min
* Clinically significant alanine transaminase (3×the upper limit of normal [ULN]) and/or bilirubin (2×ULN) values

Sex: All
Age Groups: Child, Adult, Older Adult

REFERENCES:
- See also: Sponsor website — http://taurx.com